CLINICAL TRIAL: NCT02846519
Title: An Open-Label, Single-Dose Study to Assess the Pharmacokinetics, Safety, and Tolerability of Intranasally Administered Esketamine in Healthy Han Chinese, Korean, Japanese, and Caucasian Subjects and the Effects of Rifampin on the Pharmacokinetics of Intranasally Administered Esketamine
Brief Title: Pharmacokinetic, Safety, and Tolerability Study of Intranasally Administered Esketamine in Healthy Han Chinese, Korean, Japanese, and Caucasian Participants and the Effects of Rifampin on the Pharmacokinetics of Intranasally Administered Esketamine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108128; ESKETINTRD1008 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-07-25; First posted 2016-07-27 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — Esketamine; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Esketamine (Experimental): Participants in Cohort 1 (Han Chinese participants), Cohort 2 (Korean participants) and Cohort 3 (Japanese participants ) will receive 100-microliter (mcL) spray of 14 percent (%) esketamine solution (14 milligram [mg]) into each nostril at Time 0 and 5 minutes later for a total dose of 56 milligram (mg) in Period 1.
  Interventions: Drug: Esketamine
- Esketamine+Rifampin (Experimental): Participants in Cohort 4 (Caucasian participants) will receive a 56-mg intranasal esketamine dose regimen on Day 1 in treatment period 1 followed by rifampin from Day -6 to Day -1 of treatment Period 2 and followed by 56-mg intranasal esketamine dose regimen on Day 1 in treatment period 2.
  Interventions: Drug: Esketamine; Drug: Rifampin

INTERVENTIONS:
Drug: Esketamine — 100-mcL spray of 14% esketamine solution (14 mg) for a total dose of 56 mg.
Drug: Rifampin — 2 capsules (300 mg each) of rifampin.
  Arms: Esketamine+Rifampin

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics of intranasally administered esketamine in healthy Han Chinese, Korean, Japanese, and Caucasian participants and to evaluate the effects of rifampin on the pharmacokinetics of intranasally administered esketamine in healthy Caucasian participants.

ELIGIBILITY:
Inclusion Criteria:

* For Cohort 1: healthy Han Chinese participants 20 to 55 years of age, inclusive, who have resided outside of China for no more than 10 years and have parents and maternal and paternal grandparents who are of Han Chinese ethnicity For Cohort 2: healthy Korean participants 20 to 55 years of age, inclusive, who have resided outside of Korea for no more than 10 years and have parents and maternal and paternal grandparents who are of Korean ethnicity For Cohort 3: healthy Japanese participants 20 to 55 years of age, inclusive, who have resided outside of Japan for no more than 10 years and have parents and maternal and paternal grandparents who are of Japanese ethnicity For Cohort 4: healthy Caucasian participants 20 to 55 years of age, inclusive Participants must be within +/-7 years and +/-20 percent (%) of the combined mean age and mean body weight at Screening, respectively, of Cohort 1, Cohort 2, and Cohort 3
* Body mass index (BMI; weight [kilogram]/height^2 [m]^2) between 18 and 30 kilogram per meter square (kg/m^2), inclusive, and a body weight not less than 47 kilogram (kg)
* If a woman, must have a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test at Screening
* If a woman, must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for 1 month after receiving the last dose of study drug
* Creatinine clearance more than equal to (>=)80 milliliters per minute (mL/min) based on Cockroft-Gault equation

Exclusion Criteria:

* Current significant psychiatric disorder including but not limited to psychotic, bipolar, major depressive, or anxiety disorder
* Clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at Screening or Day -1 of Period 1 as deemed appropriate by the investigator
* Clinically significant abnormal physical examination, vital signs, or 12 lead electrocardiogram (ECG) at Screening or Day -1 of Period 1 as deemed appropriate by the investigator
* History of drug or alcohol abuse disorder within the past 1 year, or a reason to believe a participant has such a history
* Regular use of intranasal tobacco powder within the past 1 year, or a reason to believe a participant has such a history

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2016-02-26 (Actual); Primary Completion 2016-05-28 (Actual); Study Completion 2016-05-28 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Up to Day 2
  The Cmax is the maximum observed plasma concentration.
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Up to Day 2
  The Tmax is defined as actual sampling time to reach maximum observed plasma concentration.
Time to Last Observed Quantifiable Plasma Concentration (Tlast) | Up to Day 2
  The Tlast is the time to last observed quantifiable plasma concentration.
Area Under the Plasma Concentration-time Curve From Time 0 to 12 Hours (AUC12h) | Up to Day 2
  The (AUC12h) is the area under the plasma concentration-time curve from time 0 to 12 hours Post-dose.
Area Under the Plasma Concentration-Time Curve From Time Zero to Time of the Last Quantifiable Concentration AUC(0-last) | Up to Day 2
  The AUC (0-last) is the area under the plasma concentration-time curve from time 0 to time of the last quantifiable concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) | Up to Day 2
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(0-last) and C(0-last)/lambda(z), wherein AUC(0-last) is the area under the plasma concentration-time curve from time 0 to time of the last quantifiable concentrations; C(0-last) is the last observed quantifiable concentration; and lambda(z) is elimination rate constant.
Elimination Half-life (t1/2) | Up to Day 2
  Elimination half-life (t [1/2]) is associated with the terminal slope (lambda [z]) of the semi logarithmic drug concentration-time curve, calculated as 0.693/lambda(z).
Rate Constant (Lambda[z]) | Up to Day 2
  Lambda(z) is first-order rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AE) as a Measure of Safety and Tolerability | Up to Follow-up (45 days)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Cypress, California, United States

REFERENCES:
- [Derived] Perez-Ruixo C, Rossenu S, Zannikos P, Nandy P, Singh J, Drevets WC, Perez-Ruixo JJ. Population Pharmacokinetics of Esketamine Nasal Spray and its Metabolite Noresketamine in Healthy Subjects and Patients with Treatment-Resistant Depression. Clin Pharmacokinet. 2021 Apr;60(4):501-516. doi: 10.1007/s40262-020-00953-4. Epub 2020 Oct 31. PMID 33128208